CLINICAL TRIAL: NCT01506661
Title: Immune Response to Varicella Zoster Vaccination (ZOSTAVAX) in Subjects With Rheumatoid Arthritis
Brief Title: Safety of Zostavax Vaccination in Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oklahoma Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OMRF11-53
Record Dates: First submitted 2012-01-05; First posted 2012-01-10 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis; Varicella Zoster
Keywords: Rheumatoid arthritis; vaccination; immune response; varicella zoster
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Herpes Zoster Vaccine; Vaccines

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rheumatoid Arthritis (Experimental): 10 subjects with mild rheumatoid arthritis aged 50 years and older will be enrolled and will receive a single dose of Zostavax vaccine.
  Interventions: Drug: Zostavax (varicella zoster virus) vaccine
- Healthy Subjects (Active Comparator): 10 healthy subjects aged 50 years or older who have not been previously immunized, will receive a single injection of Zostavax.
  Interventions: Drug: Zostavax (varicella zoster virus) vaccine

INTERVENTIONS:
Drug: Zostavax (varicella zoster virus) vaccine — Standard vaccination protocol for Zostavax will be utilized. 0.65 ml (19,400 plaque forming units) Zostavax will be administered subcutaneously once at the baseline visit

SUMMARY:
Herpes Zoster (shingles) is caused by reactivation of latent varicella zoster virus (VZV) that usually occurs decades following initial exposure. The risk of developing shingles increases with age. Shingles presents as a painful, itchy blistering rash that usually involves a single portion of the skin and lasts about 7-10 days. The risk of developing shingles increases with age in healthy people, and has been shown in some studies to be increased in people with rheumatoid arthritis and other autoimmune diseases.

Zostavax, a live-attenuated vaccine against the varicella zoster virus, was first approved by the FDA for the prevention of Shingles among people 60 years and older, and is now approved for use in people aged 50 years and older. Because rheumatoid arthritis and some of the medications used to treat rheumatoid arthritis can impair the body's immune system, it is not known how much of an immune response can be generated in people with rheumatoid arthritis.

The goals of this study are to measure the immune response after standard vaccination with Zostavax in people with rheumatoid arthritis in comparison to people with healthy immune systems. All participants will be 50 years old or older, and subjects with rheumatoid arthritis will not be eligible if they are taking certain biologic medications, including TNF inhibitors (Etanercept or Adalimumab). Ten healthy subjects and 10 subjects with rheumatoid arthritis will all receive a single vaccination with Zostavax, then will be followed for 12 weeks to assess the immune response and for the development of local rash or other potential side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Willing and able to provide written informed consent
* History of primary varicella vaccination or positive VZV IgG antibodies
* Diagnosis of RA according to ACR criteria for > 1 year, or healthy control subject
* Stable, mild disease activity as defined by a DAS28 score of 4.0
* Current medical treatment for RA has been stable for 4 weeks prior to screening
* Acceptable immunosuppressive medications are limited to Prednisone ≤ 10 mg daily Methotrexate ≤ 20 mg weekly Hydroxychloroquine ≤ 6.5 mg/kg daily Any TNF inhibitor
* Female subjects of childbearing potential and non-sterile males must agree to use acceptable form of contraception for the duration of the study

Exclusion Criteria:

* History of receiving any VZV-containing vaccine
* History of herpes zoster reactivation (shingles) within 5 years of enrollment
* Received any vaccine within 6 weeks
* Known Hepatitis B, C or HIV virus infection
* History of drug or alcohol abuse within 1 year
* Rituximab therapy within 2 years of screening
* Cyclophosphamide within 6 months of screening
* Biologic therapy: TNF inhibitors with longer half-lives (infliximab, golimumab, etc), or other non-TNF biologic therapies (IL-1 or IL-6 inhibition, or CTLA-4Ig)
* Use of mycophenolate mofetil within 3 months of screening
* History of receiving immunoglobulin or other blood product within 3 months of screening
* Allergic reaction, intolerance or other contraindication to use of famciclovir.
* Has received an experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) within 3 months of screening; or expects to receive another experimental/investigational agent within 6 months post immunization.
* Pregnant or lactating women
* Unwilling to use acceptable method of contraception for the duration of the study
* WBC <3.0; ANC <1500; CD4+ <200
* Proteinuria >1.5 mg/day
* Impaired renal function defined by serum Cr >1.5
* Transaminases > 2x upper limit of normal
* DAS28 > 4
* Anticipation of need to increase level of immunosuppression or add biologic therapy for 6 months following dosing.
* History of neoplastic disease within 5 years of screening, except for completely excised non-melanoma cancer of the skin or in-situ carcinoma of the uterine cervix.
* History of any hematological malignancy, current bleeding disorder or taking anticoagulant medication (heparin or warfarin).
* Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2017-12 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Safety and development of localized herpes zoster lesions | 12 weeks
  The primary outcome of the study is assessment of adverse events, including injection site reactions and development of zoster-like lesions, following vaccination in subjects with RA compared to healthy subjects

SECONDARY OUTCOMES:
Immunogenicity | 6 weeks
  The secondary objective of the study is immunogenicity. Specifically, the change from baseline in varicella-zoster virus-specific cell mediated immunity (assessed by IFN-g ELISpot) between subjects with RA and healthy subjects will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Chakravarty, MD, Principal Investigator — Oklahoma Medical Research Foundation
Locations (1):
- Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No